CLINICAL TRIAL: NCT06957600
Title: Navigational Bronchoscopy Versus CT-Guided Radioisotope Markings: A Randomized Controlled Trial of Preoperative Localization in Uniportal VATS Wedge Resections
Brief Title: The Comparison of Navigational Bronchoscopic and CT-Guided Preoperative Markings in Minimally Invasive Thoracic Surgery
Acronym: NaviGuide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Csaba Márton, Clinical surgeon, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMEÜ/2368-1/2022/EKU; 2025-522130-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: VATS; Lung; ICG (Indocyanine Green)
Keywords: VATS; ICG; navigational bronchoscopy; CT-guided radioisotope targeting; surgical margin; questionnaire; time
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-center, randomized clinical trial comparing navigational bronchoscopic marking using indocyanine green dye (NAVIB) with CT-guided transthoracic marking using macroalbumin-aggregated Technetium-99 (CTI). The investigators plan to enroll patients with lung nodules measuring between 1 and 3 cm of unknown origin who are undergoing wedge resections.
  In the surgical approach, the investigators exclusively utilize video-assisted techniques (VATS), and all operations in this trial are intended to be performed using a uniportal approach. This study adheres to the guidelines outlined in the Helsinki Declaration and complies with all local regulatory requirements. All participants provided informed consent before undergoing surgery. The procedures will be conducted in the Department of Thoracic Surgery at the National Institute of Oncology in Budapest, which is affiliated with Semmelweis University. All surgeries will be performed by experienced surgeons.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization occurs before surgery and is stratified by the operating surgeon using a random permuted block design with block sizes of 2 and 4. This method ensures balance among the surgeons and prevents long runs of the same group. The pathologist responsible for assessing the resections will not have access to group assignments. In this trial, only the patients, the pathologist, and the statisticians will be blinded. Due to the nature of the techniques, it is not possible to blind the surgeons and operative staff since both methods require different equipment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigational bronchoscopy (Active Comparator): For electromagnetic navigational bronchoscopic markings, the investigators use the Medtronic SuperDimension system. The process starts with a planning phase in which a thin-sliced (0.8-1.25 mm) CT scan is uploaded into the software, segmenting the airways and reconstructing the bronchial tree, allowing us to plan the best route to the lesion. During the procedure, the patient lies supine on a board emitting a low-frequency electromagnetic field. An Olympus™ bronchoscope with an extended working channel (EWC) is employed, and a locatable guide is placed into the airway. Registration matches the patient's airway to the virtual bronchial tree. Once the investigators reach the lesion, they secure the EWC and administer 2 ml of ICG 5 mg/ml solution through a 21G TBNA needle to mark it. After removing the bronchoscope, selective intubation is performed. The investigators proceed to surgery using a near-infrared Olympus optic.
  Interventions: Procedure: Preoperative marking
- CT guided markings (Active Comparator): Localization of lung lesions before surgery using CT-guided transthoracic 99mTc isotope placement (CTI) follows a specific protocol. The investigators prepare 99mTc-MAA using macroalbumin and Tc-99m, targeting 220-240 MBq in 3 ml and administering 14-16 MBq (0.2 ml) while considering the remaining syringe volume. An interventional radiologist performs the marking on the same day as the surgery, ideally in the morning. Patients are positioned for easy access to the lesion. Native CT images confirm nodule localization. Local anesthetic, typically 20 ml of 10 mg/ml Lidocaine, is injected after confirming the entry point with a 22G needle. The isotope is injected through a 15 cm 22G applicator. A final CT scan checks for complications before transferring the patient for surgery. In the operating theater, the Europrobe detects the nodule marked prior to wedge resection. Isotope marking occurs two hours before surgery, with repetition required if more than six to eight hours elapse.
  Interventions: Procedure: Preoperative marking

INTERVENTIONS:
Procedure: Preoperative marking — Applying markings prior to uniport VATS wedge resections helps localize small, potentially early-stage lung tumors. After marking, the patients are positioned laterally and receive general anesthesia with single-lung ventilation. The investigators perform VATS wedge resection using uniportal techniques. The utility incision is made in the 5th intercostal space between the anterior and mid-axillary lines. Insufflation is not typically utilized. The lesion is localized, elevated, and confirmed by palpation. The investigators then staple around the lesion using the Endo GIA™ ultra universal stapler with an Articulating Reload featuring Tri-Staple™ Technology in 45 or 60 mm lengths, choosing purple or black loads based on parenchyma thickness. Finally, the investigators close the wound and place one chest drain in the thoracic cavity, set to active suction of 5-10 cm of water.

SUMMARY:
This clinical trial aims to determine whether navigational bronchoscopic or CT-guided marking is more effective for localizing small pulmonary nodules in minimally invasive thoracic surgery. It will also assess the safety of both methods. The main questions to answer are:

* Which of the two methods enables the surgeon to locate the lesion more quickly during surgery?
* Does using the newer navigational bronchoscopic method reduce the number of insufficient resections, meaning that the lesions were not completely removed, thus affecting the surgical margin?

Researchers will compare navigational bronchoscopic ICG (visible green dye on the screen) marking to CT-guided transthoracic radioisotope targeting (a substance that emits radiation and can be detected with a specific device) to evaluate whether bronchoscopy with ICG dye is equally effective or even superior without exposing patients to radiation.

Participants will:

* Undergo an additional procedure before surgery to make the lesions detectable (Preoperative marking).
* Proceed to surgery in accordance with standard practices.
* Visit the clinic once after three weeks for follow-up checks and tests.
* Grant access to the pathological results for researchers to analyze and store data.

DETAILED DESCRIPTION:
Two different preoperative markings have proven invaluable for excising smaller pulmonary lesions. Electromagnetic navigation bronchoscopy (NAVIB) provides a more minimally invasive approach, particularly advantageous for centrally located lesions or patients with a higher risk of pneumothorax. CT-guided transthoracic radioisotope marking (CTI), on the other hand, is highly accurate for peripheral lesions and allows real-time confirmation of the marker's placement. However, it remains unclear whether one technique is superior under specific surgical conditions.

This study is a single-center, 1:1 randomized controlled trial evaluating whether NAVIB using indocyanine green dye or CTI with macroalbumin-aggregated technetium-99 99 is more effective for localization during uniportal wedge resections of lung nodules ranging from 10 to 30 mm. The primary endpoint is the duration of the surgical procedure, with secondary endpoints including complication rates, surgical margin, and surgeon satisfaction assessed through specific questionnaires.

The investigators have completed a running-up phase of the study and conducted a retrospective analysis of the data since 2022. They plan to randomize 81 patients, believing that ICG dye marking will facilitate the surgery, reduce operating time, and enhance the visibility of lung nodules. Based on preliminary data, the investigators expect an average time reduction of 10 minutes, with a standard deviation of 15 minutes. Using a power of 0.8 with a 0.05 alpha level, they determined that 74 patients are needed for the primary outcome. With an anticipated loss to follow-up or exclusions of 10%, the final target has been extended to 81 patients. Recruitment will begin once the trial has been registered internationally.

The results will be analyzed using a two-sided t-test for continuous variables (e.g., length of surgeries) and a chi-squared test for categorical variables when appropriate (e.g., complications and surgical margin positivity). In the questionnaire, the investigators will utilize a scale from 1 (not helpful) to 4 (very helpful) to assess surgeons' subjective preferences.

These results could help evaluate the safety and efficiency of both techniques, which is essential in choosing between the available marking methods and could aid in establishing new protocols.

ELIGIBILITY:
In this study, patients with lung nodules between 10 and 30 mm (under clinical IC or lower stage if it was a case of NSCLC) who are fit for surgery will be enrolled. The investigators will collect epidemiological data, including age, race, gender, Charlson Comorbidity Index, smoking history, medications taken, previous surgeries, significant diseases, BMI, and detailed parameters of the radiological size of the tumor preoperatively. Within two months before surgery, the investigators will conduct a contrast-enhanced chest CT, which will include the upper abdomen and lung function tests (FVC, FEV1, DLCO). Patients who had previous thoracic surgery, are under 18 or over 85 years of age, or have FVC or FEV1 less than 60% will be excluded. Any patient unsuitable for the complete preoperative diagnostic procedure will also be excluded (for example, where contrast material is contraindicated in chronic kidney failure). Pathological parameters of the lesion will be evaluated within four weeks after surgery. Imaging will be conducted at least during the one-month follow-up to monitor complications.

Summary:

Inclusion Criteria:

* Aged from 18 to 85
* 1-3 cm lung nodules
* planned procedure VATS uniportal diagnostic wedge

Exclusion Criteria:

* Previous thoracic surgery
* CCI greater than 12
* Long-term steroid treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Time of Surgery | From the initiation of anesthesia to the completion of the surgery
  Time needed for completion of wedge resection in minutes
Surgical Satisfaction Survey | From the completion of surgery within 24 hours
  The investigators assess the surgeons' experiences after the surgery using a questionnaire consisting of 9 questions, with answers on a scale from 1 to 4, where 1 is a poor outcome, 2 is neutral, 3 is acceptable, and 4 is a favorable outcome.
  Questions:
  1. How difficult was locating the lesion during the surgery?
  2. How challenging was the location of the lesion during the surgery?
  3. How challenging was taking out the lesion and positioning the stapler?
  4. How satisfied is the surgeon with the speed of the operation compared to the planned surgical time?
  5. After removal, did the resected specimen contain the lesion?
  6. Were there any issues with the marking? (e.g., gamma camera malfunction)
  7. How effective was the preoperative marking in helping to locate the lesion?
  8. How accurately did the marking correspond to the actual location of the lesion?
  9. How satisfied was the surgeon with the quality of the marking overall?

SECONDARY OUTCOMES:
Complication rates | From the surgery up to 4 weeks
  Postoperative complications will be assessed based on the Ottawa Thoracic Morbidity & Mortality score system, a thoracic complication scoring system that follows the principles of the Clavien-Dindo score.
Hospital stay (days) | From the surgery up to 4 weeks
  The number of days between surgery and discharge
Tube duration days | From the surgery up to 4 weeks
  The number of days after which the investigators can remove the thoracic drain.
Conversion rates | During surgery
  Conversion is defined as an anterolateral thoracotomy that is large enough to allow the surgeon's hand access to the thoracic cavity.
The length of surgical margins in mm | Within 3 weeks after surgery
  The smallest distance between the lesion and the stapling line, also referred to as the surgical margin, is measured by the pathologist and expressed in mm.
The frequency of surgical margins greater than or equal to 10 mm | From the surgery in 3 weeks
  It is considered an incomplete or suboptimal resection if the resection margins do not exceed 10 mm; it is also correlated with a higher recurrence rate. That is why the investigators create a binary variable: "yes" if the length of the surgical margin is greater than or equal to 10 mm, and "no" if it is smaller than that.

CONTACTS AND LOCATIONS:
Overall Officials: Áron Ghimessy, MD. PhD. MSc, Study Director — Semmelweis
Locations (1):
- Semmelweis University- National Institute of Oncology Department of Thoracic Surgery, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
The investigators take data control seriously. In the investigator's initial approach, the investigator does not share patients' confidential data with any third party. The primary patient consent form was created with this principle in mind. Once the study is completed and demonstrates potential benefits for scientific purposes, the investigator may consider sharing the data if requested.

REFERENCES:
- [Background] Bawaadam H, Benn BS, Colwell EM, Oka T, Krishna G. Lung Nodule Marking With ICG Dye-Soaked Coil Facilitates Localization and Delayed Surgical Resection. Ann Thorac Surg Short Rep. 2023 Feb 27;1(2):221-225. doi: 10.1016/j.atssr.2023.02.010. eCollection 2023 Jun. PMID 39790308
- [Background] Yanagiya M, Kawahara T, Ueda K, Yoshida D, Yamaguchi H, Sato M. A meta-analysis of preoperative bronchoscopic marking for pulmonary nodules. Eur J Cardiothorac Surg. 2020 Jul 1;58(1):40-50. doi: 10.1093/ejcts/ezaa050. PMID 32563193
- [Background] Lee MO, Jin SY, Lee SK, Hwang S, Kim TG, Song YG. Video-assisted thoracoscopic surgical wedge resection using multiplanar computed tomography reconstruction-fluoroscopy after CT guided microcoil localization. Thorac Cancer. 2021 Jun;12(11):1721-1725. doi: 10.1111/1759-7714.13968. Epub 2021 May 4. PMID 33943015
- [Background] Farkas A, Kocsis A, Andi J, Sinkovics I, Agocs L, Meszaros L, Torok K, Bogyo L, Radecky P, Ghimessy A, Gieszer B, Lang G, Renyi-Vamos F. [Minimally invasive resection of nonpalpable pulmonary nodules after wire- and isotope-guided localization]. Orv Hetil. 2018 Aug;159(34):1399-1404. doi: 10.1556/650.2018.31148. Hungarian. PMID 30122061
- [Background] Nelson DB, Tayob N, Mitchell KG, Correa AM, Hofstetter WL, Sepesi B, Walsh GL, Vaporciyan AA, Swisher SG, Antonoff MB, Roth JA, Rice DC, Vauthey JN, Mehran RJ. Surgical margins and risk of local recurrence after wedge resection of colorectal pulmonary metastases. J Thorac Cardiovasc Surg. 2019 Apr;157(4):1648-1655. doi: 10.1016/j.jtcvs.2018.10.156. Epub 2018 Nov 26. PMID 30635188
- [Background] Schwarz Y, Greif J, Becker HD, Ernst A, Mehta A. Real-time electromagnetic navigation bronchoscopy to peripheral lung lesions using overlaid CT images: the first human study. Chest. 2006 Apr;129(4):988-94. doi: 10.1378/chest.129.4.988. PMID 16608948
- [Background] Krauel L, Pasten A, Gorostegui M, Mane S, Martin Gimenez MP, Coronas M, Carrasco Torrents R, Mora J. Use of Radioguided Surgery for Small and Difficult-to-Locate Relapsed MIBG (+) High-Risk Neuroblastoma Lesions. Cancers (Basel). 2024 Sep 30;16(19):3348. doi: 10.3390/cancers16193348. PMID 39409967
- [Background] Galetta D, Rampinelli C, Funicelli L, Casiraghi M, Grana C, Bellomi M, Spaggiari L. Computed Tomography-Guided Percutaneous Radiotracer Localization and Resection of Indistinct/Small Pulmonary Lesions. Ann Thorac Surg. 2019 Sep;108(3):852-858. doi: 10.1016/j.athoracsur.2019.03.102. Epub 2019 May 7. PMID 31075251
- [Background] Ivanovic J, Al-Hussaini A, Al-Shehab D, Threader J, Villeneuve PJ, Ramsay T, Maziak DE, Gilbert S, Shamji FM, Sundaresan RS, Seely AJ. Evaluating the reliability and reproducibility of the Ottawa Thoracic Morbidity and Mortality classification system. Ann Thorac Surg. 2011 Feb;91(2):387-93. doi: 10.1016/j.athoracsur.2010.10.035. PMID 21256276
- [Background] Park CH, Han K, Hur J, Lee SM, Lee JW, Hwang SH, Seo JS, Lee KH, Kwon W, Kim TH, Choi BW. Comparative Effectiveness and Safety of Preoperative Lung Localization for Pulmonary Nodules: A Systematic Review and Meta-analysis. Chest. 2017 Feb;151(2):316-328. doi: 10.1016/j.chest.2016.09.017. Epub 2016 Oct 4. PMID 27717643
- [Background] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456
- [Background] Keating J, Singhal S. Novel Methods of Intraoperative Localization and Margin Assessment of Pulmonary Nodules. Semin Thorac Cardiovasc Surg. 2016 Spring;28(1):127-36. doi: 10.1053/j.semtcvs.2016.01.006. Epub 2016 Feb 4. PMID 27568150